CLINICAL TRIAL: NCT04479917
Title: A Multi-Center ,Randomized, Double-Blind, Placebo-Controlled, Dose-Exploring Study to Evaluate the Efficacy and Safety of TPN171H in China Male Patients With Erectile Dysfunction
Brief Title: Efficacy and Safety of TPN171H in the Patients With Erectile Dysfunction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vigonvita Life Sciences (Industry)
Collaborators: Shanghai Institute of Materia Medica, Chinese Academy of Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TPN171H-E201
Record Dates: First submitted 2020-07-11; First posted 2020-07-21 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2021-12

CONDITIONS: Erectile Dysfunction
Keywords: Erectile Dysfunction; TPN171H; Simmerafil
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- TPN171H 5mg group (Experimental): TPN171H 5mg tablet + Placebo 10mg 2 tablets
  Interventions: Drug: TPN171H
- TPN171H 10mg group (Experimental): TPN171H 10mg tablet + Placebo 5mg tablet+ Placebo 10mg tablet
  Interventions: Drug: TPN171H
- TPN171H 20mg group (Experimental): TPN171H 10mg 2 tablets + Placebo 5mg tablet
  Interventions: Drug: TPN171H
- Placebo group (Placebo Comparator): Placebo 5mg tablet+ Placebo 10mg 2 tablets
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: TPN171H — Pharmaceutical form;tablets Route of administration:;oral;Administered 30 minutes to 4 hours prior to initiation of sexual activity for a duration of 8 weeks to use no more than one dose in any 24-hour period
  Other Names: Simmerafil
  Arms: TPN171H 10mg group; TPN171H 20mg group; TPN171H 5mg group
Drug: placebo — Pharmaceutical form;tablets Route of administration:;oral;Administered 30 minutes to 4 hours prior to initiation of sexual activity for a duration of 8 weeks to use no more than one dose in any 24-hour period
  Arms: Placebo group

SUMMARY:
This is an exploratory clinical study to presume the optimum usage and dosage for a therapeutic confirmatory study by evaluating the efficacy and safety of TPN171H 5mg, 10mg, 20mg or placebo administered orally in patients with erectile dysfunction. In conclusions, Patients with erectile dysfunction (ED) were administered placebo, TPN171H 5mg, 10mg or 20mg 30 minutes to 4 hours before sexual intercourse for 8 weeks.

DETAILED DESCRIPTION:
This is a Phase II study in 240 ED patients, which consists of 3 part: 1) a 4-week run-in period without any ED treatment; 2)randomization to 8 weeks of treatment with TPN171H or placebo; and 3) a 1-week follow-up period for continued adverse event monitoring.

The effects of TPN171H on ED will be evaluated using the IIEF-EF and SEP diaries. The IIEF-EF will be administered at baseline and at 4-week intervals following initiation of treatment, meanwhile the SEP diary will be completed by patients after each sexual attempt throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Male patients aged ≥22 with ED, defined as an inability to achieve or maintain a penile erection sufficient for satisfactory sexual intercourse, evident for at least 3 months;
* Patients whose IIEF-EF domain score is < 26;
* Patients in a stable, heterosexual relationship for at least 3 months and during the study;
* Patients who are willing to stay away from any other medicines or treatments for ED during this study period;
* Patients who are willing to have 4 or more attempts of sexual intercourse each month, demonstrated compliance with the study protocol, including drug administration, diary completion, and scheduled study visits, during the qualifying trial;
* Patients who are willing to take proper contraceptive during the study and within 3 months after the study completed;
* Patients who have voluntarily decided to participate in this study, and signed the informed consent form.

Exclusion Criteria:

* Patients with anatomical malformations of the penis;
* Patients with primary hypoactive sexual desire;
* Patients with ED, which is caused by any other primary sexual disorder, like hypopituitarism, hypothyroidism, or hypogonadism.
* Patients with ED ,which is caused by spinal injury or have had a radical prostatectomy or other surgery ;
* Patients who have a penile implant;
* Patients who have a history of hypersensitivity to other PDE5 inhibitors or who have not responded to them;
* Patients with the following cardiovascular disease:

Myocardial infarction or stroke within the last 6 months; Unstable angina or angina occurring during sexual intercourse; New York Heart Association Class 2 or greater heart failure in the last 6 months; Uncontrolled hypotension (<90/60mmHg), or uncontrolled hypertension (≥160/95mmHg); Orthostatic hypotension.

* Patients administered with the following medications:

Nitrate/Nitric oxide (NO) donors; Androgens, anti-androgen, trazodone; Agents that significantly affect the CYP3A4 intermediary metabolism.

* Diabetic patients whose FBS is over 1.5 fold of normal value, or whose HbA1c exceeds 9%, or with diabetes complications, such as diabetic nephropathy, peripheral neuropathy;
* Patients with hepatic or renal dysfunction as per the following: AST, ALT≧2*ULN, serum creatinine exceeds 20% of the upper limit of normal value;
* Patients with active gastrointestinal ulcers and bleeding disorders;
* Patients who have a history of NAION, or with a known genetically degenerative retinopathy, including retinitis pigmentosa;
* Patients who have a history of sudden decrease or loss of hearing;
* Patient with a history of malignancy;
* Patients with a major refractory psychiatric disorder or significant neurological abnormalities;
* Patients with alcohol addiction or persistent abuse of drugs of dependence;
* Patients who are participating or discontinued participation in the past 3 months from any other clinical trial, or are planning to father a baby or are in a relationship with a pregnant partner.
* For other reasons besides the aforementioned cases, patient whose participation is deemed inappropriate due to clinically significant findings according to the medical decision of the principal investigator or the study personnel.

Min Age: 22 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2020-07-23 (Actual); Primary Completion 2021-07-26 (Actual); Study Completion 2021-07-26 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in the International Index of Erectile Function - Erectile Function Domain (IIEF-EF) at Week 8 | baseline and 8 weeks
  The primary efficacy variable was the change in the EF domain scores of the IIEF questionnaire from baseline, calculated by comparing total scores from questions 1-5 and 15 from the IIEF questionnaire .
Change From Baseline in Question 2 of the Patient Sexual Encounter Profile (SEP) Diary at Week 8 in Percentage of Yes Responses | baseline and 8 weeks
  Assessed was the mean change from baseline in the percentage of Yes responses to the SEP diary Question 2. "Were you able to insert your penis into your partner's vagina when you are trying to have sex ?" Data are presented as the mean percentage of yes responses per participant.
Change From Baseline in Question 3 of the Patient Sexual Encounter Profile (SEP) Diary at Week 8 in Percentage of Yes Responses | baseline and 8 weeks
  Assessed was the mean change from baseline in the percentage of Yes responses to the SEP diary Question 3. "Did your erection last long enough for you to have successful intercourse?" Data are presented as the mean percentage of yes responses per participant.

SECONDARY OUTCOMES:
Change From Baseline to 4 Week and 8 Week Endpoint in International Index of Erectile Function (IIEF),Orgasmic Functions | baseline ,4 weeks and 8 weeks
  Self-reported Orgasmic Functions over the past 4 weeks. Scores range from 0 (low/no satisfaction) to 5 (high satisfaction), thus the 2 questions of the IIEF-OF domain range from 0 to 10.
Change From Baseline to 4 Week and 8 Week Endpoint in International Index of Erectile Function (IIEF) ,Sexual Desire | baseline ,4 weeks and 8 weeks
  Self-reported Sexual Desire over the past 4 weeks. Scores range from 0 (low/no satisfaction to 5 (high satisfaction), thus the 2 questions of the IIEF-SD domain range from 0 to 10.
Change From Baseline to 4 Week and 8 Week Endpoint in International Index of Erectile Function (IIEF),Intercourse Satisfaction | baseline ,4 weeks and 8 weeks
  Self-reported intercourse satisfaction over the past 4 weeks. Scores range from 0 (low/no satisfaction) to 5 (high satisfaction), thus the 3 questions of the IIEF-IS domain range from 0 to 15.
Change From Baseline to 4 Week and 8 Week Endpoint in International Index of Erectile Function (IIEF), Overall Satisfaction | baseline ,4 weeks and 8 weeks
  Self-reported overall satisfaction over the past 4 weeks. Scores range from 0 (low/no satisfaction to 5 (high satisfaction), thus the 2 questions of the IIEF-OS domain range from 0 to 10.
Change From Baseline in Question 2 of the Patient Sexual Encounter Profile (SEP) Diary at Week 4 in Percentage of Yes Responses | baseline and 4 weeks
  Assessed was the mean change from baseline in the percentage of Yes responses to the SEP diary Question 2. "Were you able to insert your penis into your partner's vagina?" Data are presented as the mean percentage of yes responses per participant.
Sexual Encounter Profile (SEP) Diary, Question 3 Change From Baseline to Week 4 in Percentage of Yes Responses | baseline and 4 weeks
  Assessed was the mean change from baseline in the percentage of Yes responses to the SEP diary Question 3. "Did your erection last long enough for you to have successful intercourse?" Data are presented as the mean percentage of yes responses per participant.
Change From Baseline in the International Index of Erectile Function - Erectile Function Domain (IIEF-EF) ≥26 at Week 8 | baseline ,4 weeks and 8 weeks
  Assessed was the changes in the number of subjects whose IIEF domain score at the 8th week visit was ≥26.
Subgroup analysis based on ED severity categories: severe,0-10; moderate,11-16; mild,17-25. | baseline ,4 weeks and 8 weeks
  Subgroup analysis based on ED severity categories: severe,0-10; moderate,11-16; mild,17-25.
Subgroup analysis based on the time intervals between meal and medication. | baseline ,4 weeks and 8 weeks
  Subgroup analysis based on the time intervals between meal and medication.

CONTACTS AND LOCATIONS:
Overall Officials: Hui Jiang, MD, PhD, Principal Investigator — Peking University Third Hospital
Locations (12):
- China (12):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Guangzhou First People's Hospital, Guangzhou, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Second Affiliated Hospital of Suzhou University, Suzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jinlin
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning

IPD SHARING:
Plan to Share IPD: No